CLINICAL TRIAL: NCT06050122
Title: A Multicenter, Randomized, Double Blind, Vehicle-controlled, Phase 3 Efficacy and Safety Study of Patidegib Gel 2% for the Reduction of Disease Burden of Persistently Developing Basal Cell Carcinomas (BCCs) in Subjects With Gorlin Syndrome
Brief Title: Efficacy and Safety of Patidegib Gel 2% for Preventing Basal Cell Carcinomas on the Face of Adults With Gorlin Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SGT-610-01; 2023-507528-21-00 (Other: EU CT)
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Gorlin Syndrome
MeSH Terms: conditions — Basal Cell Nevus Syndrome | interventions — IPI-926

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patidegib Gel 2% (Experimental): Patidegib Gel 2% (w/w), applied topically to the face twice daily for 12 months
  Interventions: Drug: Patidegib Topical Gel
- Vehicle Gel (Placebo Comparator): Vehicle Gel, applied topically to the face twice daily for 12 months
  Interventions: Drug: Patidegib Topical Gel with no active patidegib

INTERVENTIONS:
Drug: Patidegib Topical Gel — Patidegib Gel 2% is a smooth, clear, colorless-to-yellow, viscous, hydro-alcoholic gel for topical administration.
  Other Names: Patidegib; IPI-926; Saridegib; SGT-610
  Arms: Patidegib Gel 2%
Drug: Patidegib Topical Gel with no active patidegib — Vehicle Gel consists of the excipients of Patidegib Gel with no active patidegib. It is a smooth viscous gel for topical administration.
  Other Names: Vehicle Gel; Placebo
  Arms: Vehicle Gel

SUMMARY:
The aim of this clinical study is to find out how well Patidegib Gel 2% works in preventing new basal cell carcinomas (BCCs) developing on the face of adults with Gorlin syndrome, and how safe Patidegib Gel 2% is to use.

People who take part will apply either Patidegib Gel 2% or a Vehicle Gel (with no active drug substance) to their face twice a day for a year (12 months). The number of new BCCs on the face will be compared between those who used Patidegib Gel 2% or Vehicle Gel after 12 months.

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, stratified, vehicle-controlled study of the efficacy and safety of Patidegib Gel 2%, applied topically twice daily to the face of adult subjects with Gorlin syndrome.

Subjects will be randomized (1:1) to receive either Patidegib Gel 2% or Vehicle Gel for 12 months.

The assignment of subjects to the 2 groups will be stratified by sex assigned at birth, age (≥60 or <60 years), and number of BCC lesions at the treatment area (face) (10-15, 16-30 or >30) at Baseline.

All suspicious lesions will be imaged and tracked consistently throughout the study so that new BCCs that arise can be readily identified. New BCCs will be confirmed by dermoscopic analysis through the study. The BCC images will be reviewed and assessed by a Central Photo Review Board (CPRB).

ELIGIBILITY:
Key Inclusion Criteria:

1. The subject must be at least 18 years old at the Screening Visit.
2. The subject must be confirmed to have a PTCH1 mutation.
3. The subject must have at least 10 BCCs on the face at Randomization (Baseline/Day 1).
4. The subject must be willing to abstain from application of any non-study topical medication (prescription or over the counter) to their facial skin for the duration of the trial, except as prescribed by the investigator.

Key Exclusion Criteria:

1. The subject has used topical treatment to the face or systemic therapies that might interfere with the evaluation of the study Investigational Product (IP).
2. The subject is known to have hypersensitivity to any of the ingredients in the IP formulation.
3. The subject has uncontrolled systemic disease.
4. The subject has been treated for invasive cancer within the past 5 years excluding chronic lymphocytic leukemia Stage 0, non-melanoma skin cancer, successfully treated melanoma in situ and Stage I melanoma, Stage I cervical cancer, or ductal carcinoma in situ of the breast.
5. Inefficacy of previous Hedgehog inhibitor therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of new BCCs on the face at Month 12 | Month 12
  New BCCs at Month 12 after twice-daily treatment with either Patidegib Gel 2% or Vehicle Gel for 12 months, as assessed by the CPRB

CONTACTS AND LOCATIONS:
Locations (40):
- United States (24):
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - Center for Dermatology Clinical Research, Fremont, California
  - University of California Los Angeles (UCLA) - Center for Inflammatory Bowel Diseases - Westwood Location, Los Angeles, California
  - The Dermatology Center of Newport, Newport Beach, California
  - Stanford University - Lucille Packard's Children's Hospital, Redwood City, California
  - Yale University, New Haven, Connecticut
  - Dermatology Associates of Tallahassee, Tallahassee, Florida
  - University of South Florida Health, Tampa, Florida
  - The University of Chicago Medicine, Chicago, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Health - Michigan Medicine - University Hospital, Ann Arbor, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Schweiger Dermatology P.C., Verona, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Health System, Durham, North Carolina
  - Apex Clinical Research Center, Canton, Ohio
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - SSM Health Dermatology, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - North Texas Center for Clinical Research, Frisco, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- France (3):
  - Hopital Avicenne, Bobigny
  - Centre Hospitalier Universitaire De Nantes, Nantes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (3):
  - Ludwig-Maximilians-Universitaet Muenchen (LMU) - Klinik und Poliklinik fuer Dermatologie und Allergologie, Munich, Bavaria
  - Charité Universitätsmedizin Berlin - Campus Charité Mitte, Berlin
  - DRK Gemeinnützige Krankenhaus GmbH Sachsen, Chemnitz
- Italy (3):
  - ASST Spedali Civili di Brescia, Brescia
  - AOU Maggiore della Carita, Novara
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Maastricht University Medical Center, Maastricht, Netherlands
- Spain (3):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitartio 12 De Octubre, Madrid
- United Kingdom (3):
  - The University of Birmingham, Birmingham
  - Barts Health NHS Trust - The Royal London Hospital, London
  - Northern Care Alliance NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No